CLINICAL TRIAL: NCT05209542
Title: Hysterosalpingo-Foam Ultrasonography Combined With Power Doppler, Compared With Laparoscopy in Tubal Patency Assessment in Cases of Infertility, (a Cross-sectional Study).
Brief Title: Hysterosalpingo-Foam Ultrasonography Combined With Power Doppler, Compared With Laparoscopy in Tubal Patency Assessment in Cases of Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 63
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Infertility of Tubal Origin
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysterosalpingo-Foam Ultrasonography (Active Comparator): 3-5 ml of foam contrast is to be introduced slowly into the endometrial cavity while the flow of contrast medium in each tube is evaluated using grayscale and power Doppler imaging
  Interventions: Procedure: Hysterosalpingo-Foam Ultrasonography; Procedure: Laparoscopy
- laparoscopy (Active Comparator): • Standard laparoscopic evaluation with the dye test (methylene blue staining) is to be performed 1 day after ultrasound tests with 1 day of hospitalization under general anesthesia
  Interventions: Procedure: Hysterosalpingo-Foam Ultrasonography; Procedure: Laparoscopy

INTERVENTIONS:
Procedure: Hysterosalpingo-Foam Ultrasonography — * Initial 3-5 ml of foam contrast is to be introduced slowly into the endometrial cavity while the flow of contrast medium in each tube is evaluated using grayscale and power Doppler imaging
  * Power Doppler is very helpful to confirm the direction of the flow as well as the acceleration during injection
Procedure: Laparoscopy — • Standard laparoscopic evaluation with the dye test (methylene blue staining) is to be performed 1 day after ultrasound tests with 1 day of hospitalization under general anesthesia

SUMMARY:
Women presenting with primary or secondary infertility and are undergoing investigation of tubal patency assessment will be subjected to:

* The examination is performed between days 5 and 10 of the menstrual cycle.
* Routine antibiotic prophylaxis using oral Azithromycin the day before and routine administration of NSAID rectal suppository one hour before the procedure
* Initially, real-time 2D +/- 3D vaginal ultrasound assessment of the pelvis
* The cervix is to be visualized with a Cusco speculum and to be cleaned with an antiseptic then A No. 5 pediatric Foley catheter will be introduced into the cervical os, using a tenaculum if necessary. The balloon is to be positioned in the lower uterine cavity and to be inflated with 2 ml of saline to prevent backflow of contrast medium through the cervix then the speculum will be removed and the vaginal transducer is going to be reintroduced in the longitudinal plane to confirm correct placement of the catheter.
* Initial 3-5 ml of foam contrast is to be introduced slowly into the endometrial cavity while the flow of contrast medium in each tube is evaluated using grayscale and power Doppler imaging
* Power Doppler is very helpful to confirm the direction of the flow as well as the acceleration during injection.
* Tubal patency and quality of visualization are classified according the following parameters:

  1. Flow over the whole length of the tube, fimbrial outflow or peritoneal spillage of contrast provided definite evidence of complete (i.e. proximal and distal) tubal patency.
  2. Paracornual flow only without visualization of fimbrial outflow or peritoneal spillage suggests at least proximal patency.
  3. Contrast filling of the endometrial cavity without cornual flow suggests possible tubal occlusion.
  4. Technical difficulty making tubal evaluation impossible
* Standard laparoscopic evaluation with the dye test (methylene blue staining) is to be performed 1 day after ultrasound tests with 1 day of hospitalization under general anesthesia.

DETAILED DESCRIPTION:
Women in the reproductive age group between 20 and 40 years old presenting with primary or secondary infertility ( either unexplained or suspected tubal factor by history taking ) and are undergoing investigation of tubal patency assessment

Each patient in this study will be subjected to:

* The examination is performed between days 5 and 10 of the menstrual cycle, the patient in gynecological position, preferably with the aid of one assistant.
* Routine antibiotic prophylaxis using oral Azithromycin the day before and routine administration of NSAID rectal suppository one hour before the procedure
* Initially, real-time 2D +/- 3D vaginal ultrasound assessment of the pelvic organs is to be performed using Samsung Elite with endovaginal probe of frequency 6-12 MHz
* The cervix is to be visualized with a Cussco speculum and to be cleaned with an antiseptic then A No. 5 pediatric Foley catheter will be introduced into the cervical os, using a tenaculum if necessary. The balloon is to be positioned in the lower uterine cavity and to be inflated with 2 ml of saline to prevent backflow of contrast medium through the cervix then the speculum will be removed and the vaginal transducer is going to be reintroduced in the longitudinal plane to confirm correct placement of the catheter.
* The foam contrast agent is created by combining 3-4mL of 2% lidocaine gel 12-13mL of saline and 3mL air.
* The assistant creates the foam immediately before application, moving the mixture between two connected 20-mL syringes, until a whitish suspension is obtained (approximately 10-20 times).
* Initial 3-5 ml of foam contrast is to be introduced slowly into the endometrial cavity while the flow of contrast medium in each tube is evaluated using grayscale and power Doppler imaging
* Power Doppler is very helpful to confirm the direction of the flow as well as the acceleration during injection.
* Acquisition without Doppler usually takes less than 5 s, while acquisition with power Doppler is longer(approximately 10 s)
* After dataset acquisition, Images will be stored as 2D still images, 2D clips +/- 3D volumes. the patient is to be discharged and final diagnosis is made based on the real-time observations and, if available, offline analyses of acquired datasets.
* Tubal patency and quality of visualization are classified according the following parameters:

  1. Flow over the whole length of the tube, fimbrial outflow or peritoneal spillage of contrast provided definite evidence of complete (i.e. proximal and distal) tubal patency.
  2. Paracornual flow only without visualization of fimbrial outflow or peritoneal spillage suggests at least proximal patency.
  3. Contrast filling of the endometrial cavity without cornual flow suggests possible tubal occlusion.
  4. Technical difficulty making tubal evaluation impossible e.g. absent filling of the endometrial cavity due to backflow of contrast, inability to introduce the catheter into the cervical os or maintain the catheter in the correct position preventing instillation of contrast into the endometrial cavity.
* Standard laparoscopic evaluation with the dye test (methylene blue staining) is to be performed 1 day after ultrasound tests with 1 day of hospitalization under general anesthesia.
* The raters are to be blinded to the results of the ultrasound examination until endoscopic diagnosis is to be performed
* Comparison between the results of the above mentioned techniques will be done and statistical analysis of the results will be carried out

ELIGIBILITY:
Inclusion Criteria:

Sexually active women in the reproductive age group between 20 and 40 years

* History of primary or secondary infertility ( either unexplained or suspected tubal factor by history taking )
* Tubal factor has not been investigated before or has been investigated with inconclusive results

Exclusion Criteria:

* Age less than 20 or above 40 years.
* Using contraception.
* Undiagnosed pregnancy.
* known allergy to lidocaine.
* active pelvic inflammatory disease or genital tract bleeding.
* Patent both tubes as assessed previously ( no need for exposure to further Investigation.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 119 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2021-04-03 (Actual)

PRIMARY OUTCOMES:
Tubal patency | During the ultrasound
  To evaluate the accuracy of Hysterosalpingo-Foam Sonography combined with Power Doppler in assessment of tubal patency in infertile women

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Maged M ElGoly, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided